CLINICAL TRIAL: NCT05234086
Title: Randomized, Controlled Phase II Clinical Study to Evaluate Superiority of "InbioDerm+C" Autologous Stem Cell-Based Therapy Plus Advanced Healing Compared With Advanced Healing in Diabetic Foot Ulcer Patients
Brief Title: Cell Therapy for Diabetic Foot Ulcer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto para el Desarrollo Biotecnológico y la Innovación S.A. (Other)
Collaborators: Corporación de Fomento de la Producción, Chile (Unknown)
Responsible Party: Principal Investigator, Soledad Herrera, Regulatory Affairs - Inbiocriotec, Instituto para el Desarrollo Biotecnológico y la Innovación S.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INBIO EC 201903
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Foot Ulcer Associated With Type II Diabetes Mellitus; Wound Heal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will evaluate encrypted images and tables containing healing valoration data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Healing (Active Comparator): Activities related to wound washing, microbiological load control, care of peri-ulcer tissue and application of wound healing products in accordance to condition of the ulcer
  Interventions: Procedure: Advanced healing
- InbioDerm + C plus advanced healing (Experimental): For patient who are assigned treatment with InbioDerm+C plus advanced healing a section of skin tissue and peripheral venous blood will be taken. From the skin section and through an enzymatic process with cell proliferation, skin cells will be obtained that will be integrated into de the InbioDerm+C, then will be apply to the patients with the advanced wound healing every fourteen days in accordance application program.
  Interventions: Combination Product: InbioDerm + C plus advanced healing

INTERVENTIONS:
Combination Product: InbioDerm + C plus advanced healing — For patients who are assigned to experimental treatment with InbioDerm+C plus advanced healing a section of skin tissue and peripheral venous blood will be taken. From the skin section, through an enzymatic process and cell proliferation for a period of approximately fourteen days, the cells that are integrated in the InbioDerm+C will be obtained and used to treat the foot ulcer.
  Arms: InbioDerm + C plus advanced healing
Procedure: Advanced healing — Patients who are assigned to active comparator correspond to the control treatment, which will be received advanced healing.
  Arms: Advanced Healing

SUMMARY:
Diabetes is a highly prevalent chronic disease that affects a large part of the world's population. Among the most costly complications is the diabetic foot ulcer, where its decompensation can result in limb amputation, a risk 10 to 20 times more frequent for diabetic population. Two underlying pathophysiological mechanisms are mainly identified: neuropathy and problems associated with vasculature and blood supply, in addition to the incidence of infections, which further impairs prognosis. Skin regeneration involves several overlapping and consecutive stages, which in the case of a diabetic patient are altered.

Although healing protocols have been significantly improved at the country level, and there is also a large amount of medical supplies for treatment of these wounds, there are still patients with ulcers refractory to this care that end in amputation. In response to this, new treatments have emerged that use biomaterials and cells of the patient himself, which attempt to emulate the architecture and functionality of normal tissue. Cell therapy has gained strength in recent years, with more and more studies indicating the positive effect of cell application on healing of chronic wounds with underlying pathologies, such as diabetes.

The product to be evaluated corresponds to a combined medical device, which conveys a cellular therapy, known as InbioDerm+C. The purpose of this Phase II clinical study is to determine whether InbioDerm+C treatment plus advanced healing is equal to or superior to advanced healing in a diabetic population with Wagner II grade foot ulcer treated in Villa Alemana primary care family centers, Las Américas, Juan Bautista Bravo Vega and Eduardo Frei.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old and under 75 years old.
* Patient diagnosed with DM type II.
* Patient with negative pregnancy test.
* Ulcer size with area between 1 cm2 and 12 cm2.
* Ulcer with Wagner grade II classification with less than 50% slough and no tendon exposure, validated by an external specialist after ulcer debridement.
* Ulcer age ≥ at one month.
* Patients with palpable posterior tibial and pedial pulse

Exclusion Criteria:

* Patients with non-diabetic ulcers.
* Toe ulcers.
* Patient with grade IV and V renal insufficiency.
* Pregnant or breastfeeding women, or those who are planning to conceive children.
* Clinical evidence of infection.
* Any condition or circumstance that might interfere with adherence to the treatment regimen (compliance with scheduled visits, psychiatric disorders, or drug and/or alcohol abuse)
* History of hepatitis B or hepatitis C and HIV (by internal laboratory biosafety protocols)
* Allergy to penicillin, streptomycin, and gentamicin
* Subjects undergoing treatment with immunosuppressants and corticoids.
* Subjects on anticoagulant treatment with acenocoumarol and warfarin.
* Having received any experimental treatment in the last three months (drug, biological product, medical device or cell therapy), except for the use of vaccines administered against COVID-19 (e.g. mRNA technologies, viral vector or inactivated virus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with completely closed ulcers | 16 weeks
  The principal investigation and external evaluator will assess every fifteen days the wound closure status.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Ahumada, Principal Investigator — Centro de Salud Familiar Villa Alemana
Locations (1):
- Centro de Salud Familiar de Villa Alemana, Villa Alemana, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No